CLINICAL TRIAL: NCT05756114
Title: Self Management and Recovery Training (SMART) Recovery Involvement and Alcohol Use Outcomes
Brief Title: Self Management and Recovery Training (SMART) Recovery Study
Acronym: SMART
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The focus of the project has shifted.
Sponsor: Yale University (Other)
Collaborators: Society of Addiction Psychology (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000034747
Record Dates: First submitted 2023-02-22; First posted 2023-03-06 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Self-Help Groups

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychoeducation Condition (Active Comparator): Participants receive a weekly email with a Qualtrics survey link containing psychoeducational content.
  Interventions: Other: Psychoeducational Email
- Support Group Condition (Experimental): Participants will attend six weekly online SMART Recovery meetings in groups of five to eight.
  Interventions: Behavioral: Support Group

INTERVENTIONS:
Behavioral: Support Group — Support Group condition, meetings will be held online via HIPAA-compliant Zoom and run by a trained SMART Recovery meeting facilitator
  Arms: Support Group Condition
Other: Psychoeducational Email — Participants receive a weekly email with a Qualtrics survey link containing psychoeducational content.
  Arms: Psychoeducation Condition

SUMMARY:
This study identifies whether and how online support groups may work to confer therapeutic benefits onto its participants.

DETAILED DESCRIPTION:
Online support groups (e.g., SMART Recovery) are an increasingly common non-professional intervention for people who engage in problematic alcohol use, but it is unclear how they help participants reduce their use.

The primary objective of this study is to determine whether alcohol use decreases more after attending online SMART Recovery psychoeducational support group meetings, as compared to receiving psychoeducational content alone.

The secondary objectives are to identify whether variables such as quality of life and recovery capital (i.e., resources to support recovery from addiction) relate to treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Is fluent in English and have a 6th grade reading level or higher
* AUDIT score of ≥8
* Has some desire to cut down or quit their alcohol use
* Has access to a phone or computer with reliable internet connection, a functional microphone and camera
* Is willing to consent to being audio and video recorded during the meetings

Exclusion Criteria:

* Is not able to commit to the 6 weeks of intervention and the one- and three-month follow-up.
* Has vulnerable population status (e.g., pregnant people, prisoners)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Change in past-month alcohol use: drinking days | Baseline, 1 month and 3 months
  Timeline Follow-back (TLFB) will be used via survey to characterize changes in alcohol and other drug use for study participants. Percent Drinking Days will be derived from self-report on TLFB.
Change in past-month alcohol drug use: heavy drinking days | Baseline, 1 month and 3 months
  Timeline Follow-back (TLFB) will be used via survey to characterize changes in alcohol and other drug use for study participants. Percent Heavy Drinking Days will be derived from self-report on TLFB.

SECONDARY OUTCOMES:
Change in Quality of Life | Baseline, 1 month and 3 months
  Quality of life will be assessed using the WHOQOL-BREF via survey; a 26-item self-report measure of quality of life in four domains. Scores range from 1-5. Each domain score is averaged. Higher scores indicate higher quality of life. .
Change in recovery capital | Baseline, 1 month and 3 months
  Recovery capital will be assessed using the Assessment of Recovery Capital via survey; A 50-item self-report measure of recovery capital with ten domains; each item is rated in binary, score ranges from 0-50; higher scores indicate higher recovery capital.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Potenza, PhD, MD, Principal Investigator — Yale University: Professor of Psychiatry, in the Child Study Center and of Neuroscience

IPD SHARING:
Plan to Share IPD: No